CLINICAL TRIAL: NCT02986009
Title: Be Good Parents (Parent Education)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: International Social Service Hong Kong Branch (Unknown)
Responsible Party: Principal Investigator, Nancy Xiaonan Yu, Assistant Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Parenting
Keywords: emotion management; positive and negative affect; satisfaction with parent-child relationship; subjective happiness; family harmony
MeSH Terms: interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting (Experimental): To receive the parenting intervention
  Interventions: Behavioral: Parenting
- Information (Experimental): To receive the information intervention
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Parenting — The parenting intervention consists of four weekly sessions, each lasting two hours. The intervention was designed according to the parenting characteristics of Chinese parents in Hong Kong. The four sessions cover: 1) response modification ("stop and rest"), 2) relaxation/enhancing positive moods ("relax and play"), 3) cognitive reframing ("think"), and 4) using social support ("talk and share). Discussion, practice, and questions are involved in each session.
  Arms: Parenting
Behavioral: Information — The information intervention consists of four weekly sessions, each lasting for two hours. The contents cover information and resources about education, medical care, housing, employment, and community facilities available in Hong Kong and Mainland China.
  Arms: Information

SUMMARY:
The collaborator has its vision as "To have children, individuals, families and migrants across countries live in dignity and harmony, and be contributing members to a just, humane and caring society." Parents are very significant in the families as they need nurturing, discipline, teaching, monitoring, and managing their children as well as their families. Capable and competent parents bring good child outcome and happy family. The investigators planned to serve targeted parents in two areas as 1. Emotion management and 2. Information on community resource. In the first set, the participants are expected to improve their emotion management leading to a more effective parenting. In the second set, the participants would acquire more information that enables them to better use the community resources.

To work closely with the collaborator, and based on the previous results of an effective parenting intervention, the investigators will modify the intervention to tailor the needs of targeted parents. The objectives are:

1. After completing the parenting intervention, 150 participants will, 1.1. To increase participants' emotion management strategies by 20%, 1.2. To enhance positive affect by 10%, 1.3. To decrease negative affect by 10%, 1.4. To enhance satisfaction with the parent-child relationship by 10%, 1.5. To increase subjective happiness by 8%, 1.6. To enhance family harmony by 5%, These levels of positive effects of the program were projected from the investigators' published findings.
2. After joining the information sessions about education, health care, housing, employment, and community facilities, another 150 participants will, 2.1 To know more information of Hong Kong by 50%, 2.2 To know more information of Mainland China by 50%, 2.3 To use more community resources either in Hong Kong or Mainland China by 50%.

To study the effectiveness of parenting intervention, the investigators proposed to use a randomized controlled trial (RCT) that is a type of scientific study to reduce bias. Participants in this project will be randomly allocated to either the emotional management group or the information group. As the information group has no focus on parenting, participants would show no significant improvement in emotion management strategies or satisfaction with the parent-child relationship, etc. Meanwhile, participants in the parenting intervention would show no significant improvement in knowledge about either Hong Kong or Mainland China.

DETAILED DESCRIPTION:
Parenting not only acts as an important drive for child development, also serves as one of the key determinants for family relationships. Emotion management is the essence of parenting competence. Anger, fear, joy, distress and enthusiasm are involved in the parenting process. Negative emotions of parents are associated with child abuse; while positive emotions are related to warm parenting, and promote children's early attachment with parents. In addition, parental negative emotion consistently predicts behavior problems of children. For example, children who are exposed to higher levels of maternal negative feelings, such as anger, have more difficulty regulating their own negative feelings and have greater difficulty getting along with others.

Emotion management training has been shown effective in improving parenting skills, promoting parent-child interaction, and preventing child abuse. For example, parents who attended anger control workshops reported less unrealistic expectations for their children, fewer conflicts with children, and less domestic violence toward spouse and children. However, these interventions were tested in Western culture where there is much less emphasis on academic performance of children. In addition, such interventions usually contain complex content and last for months.

The investigators developed a parenting intervention tailored for Chinese parents and reported its effectiveness in a randomized controlled trial. In this empirical study, 412 Hong Kong mothers of children aged 6 to 8 years old were randomized into the parenting arm or the control arm. The results showed that the parenting arm reported greater increase in the use of emotion management found that it was effective in increasing emotion management skills and enhancing the parent-child relationship. Participants in the parenting arm also reported lower negative affect, and higher positive affect, satisfaction with the parent-child relationship, and family harmony, compared to the control arm. The investigators' findings provide evidence for a sustainable, preventive, culturally appropriate, and cognitive behavioral-based parenting program in the community population. Considering unique dynamics of cross-boundary and new arrival families, a short and simple intervention on emotion management would benefit these parents to perform better parenting. Therefore based on the investigators' promising findings in the community setting, this proposed program aim to modify this parenting program to the needs of parents of the cross-boundary and new arrival children.

ELIGIBILITY:
Inclusion Criteria:

* The parents of cross-boundary and new arrival children whose children born or moved to Hong Kong with the one-way exit permits.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Frequency of emotion management strategies as assessed by 10 self-developed items | 1 month
  Example items include "stop thinking about the situation and do something else", "relax to calm down", "think of the reasons for child's behavior", "talk to family or friends", and "manage anger when child misbehaves"

SECONDARY OUTCOMES:
Positive and negative affect as assessed by 10 items from the Positive and Negative Affect Schedule | 1 month
Satisfaction with parent-child relationship as assessed by a single item from the Kansas Marital Satisfaction Scale | 1 month
Subjective happiness as assessed by four-item Subjective Happiness Scale | 1 month
Family harmony as assessed by Generic Family Harmony Scale | 1 month
Knowledge of Hong Kong as assessed by 20 self-developed questions | 1 month
  Examples of items are "free education is available for nine years in Hong Kong" and "Persons who have immigrated to Hong Kong less than seven years ago are not eligible to apply for public housing"

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Xiaonan Yu, Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No